CLINICAL TRIAL: NCT01902212
Title: Evaluation of an Oral Nutrition Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: BL16
Record Dates: First submitted 2013-07-03; First posted 2013-07-18 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Gastrointestinal Tolerance
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oral Nutritional Supplement (Experimental): 2 servings a day
  Interventions: Other: Oral Nutritional Supplement

INTERVENTIONS:
Other: Oral Nutritional Supplement

SUMMARY:
The objective of this study is to capture gastrointestinal tolerance (GI) information on a nutrient dense oral nutritional supplement (ONS) in healthy elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible for the study if they meet all of the following inclusion criteria:

* Male or female ≥ 60 and ≤ 90 years of age.
* Body Mass Index (BMI) > 20 but < 35.

Exclusion Criteria:

Subjects will be excluded from the study if they meet any of the following criteria:

* History of diabetes
* Antibiotic use within 1 week prior to enrollment
* Undergone major surgery less than 3 months prior to enrollment.
* Current active malignant disease or was treated within the last 6 months for cancer.
* Immunodeficiency disorder.
* Myocardial infarction within the last 3 months.
* Chronic obstructive pulmonary disease (COPD).
* Allergy to any of the ingredients in the study product.
* Obstruction of the gastrointestinal tract or other major gastrointestinal disease.
* Dementia, brain metastases, eating disorders, history of significant neurological or psychiatric disorder.
* Unintentional weight loss or weight gain ≥ 5% in last 4 weeks.
* Taking medications/dietary supplements/substances that could profoundly modulate metabolism or affect GI motility.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Gastro-Intestinal Tolerance | Study Day (SD) 1-8
  Subject questionnaire

SECONDARY OUTCOMES:
ONS Consumption | SD 1-8
  Consumption Record
Weight | Screening and SD 8

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Nelson, PhD, Study Chair — Abbott Nutrition
Locations (1):
- Biofortis Sas, Saint-Herblain, France